CLINICAL TRIAL: NCT02415322
Title: A Prospective Cohort Study to Identify Pathogenesis and Risk Factors on Internet Game and Smart Phone Addiction
Brief Title: Cohort Study on Internet Game and Smart Phone Addiction
Status: Completed | Type: Observational
Sponsor: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Hyeon Woo Yim, Professor, National Clinical Research Coordination Center, Seoul, Korea
Other Study IDs: ICURE
Record Dates: First submitted 2015-04-02; First posted 2015-04-14 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Adolescent Problems; Addictive Behavior
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: refer to mental health specialists — children who have diagnosed internet and/or smartphone disorder by psychiatrists referred to mental health specialists

SUMMARY:
The aim of this cohort study is to observe the prevalence, incidence, relapse, and remission rates of online and/or smartphone game addiction among elementary and secondary school students in Korea. In addition the investigators are going to identify risk and protective factors, to determine whether online and/or smart phone game addiction is a primary or secondary problem, and to identify outcomes for individuals who become or stop being online and smart phone game addiction.

DETAILED DESCRIPTION:
Participants:

Total 3,000 children will be enrolled the cohort and followed up for 4 years.

Procedures:

These students will be surveyed annually between 2015 and 2019. Surveys were conducted in classrooms by trained interviewer who had been trained by the research team assisted by the teachers.

Measurements

* usage and frequency of internet, internet game, and smartphone game etc.
* interpersional relationship; with family members, peer group, and teacher etc.
* personal characteristics; self esteem, social support, depression, anxiety, hyperactivity etc.
* Socio-demographic factors

ELIGIBILITY:
Inclusion Criteria:

* 3rd, 4th, and 7th grade students of selected 15 elementary and secondary schools who provide consent both the students and their parents

Exclusion Criteria:

* does not provide consent

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Tatal 3,000 elementaty and sencondary school students
Sampling Method: Non-Probability Sample
Enrollment: 2319 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
prevalence, incidence, relapse, and remission of internet gaming addiction, internet addiction, and smartphone addiction | 2-year followup point

SECONDARY OUTCOMES:
depression, anxiety, attention deficit hyperactivity disorder, suicidality prevalence, incidence, relapse, and remission rate of internet gaming, internet, and smartphone addiction | 2-year follow-up point and 4-year followup point

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Woo Yim, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jo SJ, Yim HW, Jeong H, Lee HK. Moderating Effects of Depressive Symptoms and Self-Control Trait on the Association Between Problematic Internet Gaming and Time Spent. Cyberpsychol Behav Soc Netw. 2022 Apr;25(4):237-244. doi: 10.1089/cyber.2021.0221. Epub 2022 Apr 1. PMID 35363564
- [Derived] Jeong H, Yim HW, Lee SY, Lee HK, Potenza MN, Shin Y. Preschool Exposure to Online Games and Internet Gaming Disorder in Adolescents: A Cohort Study. Front Pediatr. 2021 Nov 23;9:760348. doi: 10.3389/fped.2021.760348. eCollection 2021. PMID 34888270
- [Derived] Jeong H, Yim HW, Jo SJ, Lee SY, Lee HK, Gentile DA, Son HJ, Han HH, Kweon YS, Bhang SY, Choi JS. Gaming patterns and related symptoms in adolescents using cluster analysis: Baseline results from the Internet User Cohort for Unbiased Recognition of Gaming Disorder in Early Adolescence (iCURE) study. Environ Res. 2020 Mar;182:109105. doi: 10.1016/j.envres.2019.109105. Epub 2019 Dec 31. PMID 32069759
- [Derived] Jeong H, Yim HW, Jo SJ, Lee SY, Kim E, Son HJ, Han HH, Lee HK, Kweon YS, Bhang SY, Choi JS, Kim BN, Gentile DA, Potenza MN. Study protocol of the internet user Cohort for Unbiased Recognition of gaming disorder in Early adolescence (iCURE), Korea, 2015-2019. BMJ Open. 2017 Oct 5;7(10):e018350. doi: 10.1136/bmjopen-2017-018350. PMID 28982839